CLINICAL TRIAL: NCT02299895
Title: Professionals' Perspectives on Facilitating and Hindering Factors of Implementing Health Promotion Programs in Organizational Settings: a Qualitative Comparative Study in Austria
Brief Title: Professionals' Perspectives on Facilitating and Hindering Factors of Implementing Health Promotion Programs in Organizational Settings
Acronym: SCS
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Ludwig Boltzmann Gesellschaft (Other)
Collaborators: Ludwig Boltzmann Institut Health Promotion Research (Unknown)
Responsible Party: Principal Investigator, Wolfgang Dür, PD Dr., Ludwig Boltzmann Gesellschaft
Other Study IDs: LBG:1554
Record Dates: First submitted 2014-11-13; First posted 2014-11-24 (Estimated); Last update posted 2014-11-24 (Estimated); Status verified 2014-11

CONDITIONS: Health Promotion; Organizations
Keywords: setting approach; health promotion; organization; implementation research; qualitative study; comparison

STUDY DESIGN:
Time Perspective: Retrospective

SUMMARY:
Background:

In the field of health promotion, the 'setting approach' has gained increased attention over the last decades. Following this approach, organizations and governments are urged to invest in health and health promotion. However, the dissatisfaction with the broad definition of the term 'setting' has grown. As many health promotion programs are carried out in organizational settings, substantial work has been done on how to acknowledge organizational factors in designing and implementing health promotion programs. Organizational settings differ from others because they can also address their clients as beneficiaries of health promotion programs, also known as 'client-oriented health promotion'. Among the most prominent organizational settings for health promotion are schools and hospitals, and more recently, long-term care (LTC-) facilities. However, dissemination and implementation of client-oriented health promotion in organizational settings seem to be very challenging. Most approaches dealing with barriers to health promotion implementation in schools, hospitals, and LTC-facilities rarely reflect the specific organizational characteristics. This negligence constitutes both, a research gap in the setting approach and in the design of health promotion practice. Hence, the aim of this study is to explore professionals' (teachers', health professionals', care aids') views and attitudes that influence the implementation of client-oriented health promotion programs between schools, hospitals, and LTC-facilities in Austria.

Methods:

With that aim in mind, the investigators chose a comparative qualitative design. Semi-structured interviews will be conducted with 90 professionals (30 in schools, 30 in hospitals, and 30 in LTC-facilities). In addition, non-participant observations as well as an extensive document analysis in each setting will be undertaken. The data will be analyzed by thematic analysis. Comparisons within as well as between the organizational settings will be conducted using selected categories.

Discussion:

To date, this study is the first of its kind that compares results of individual semi-structured interviews between different organizational settings. This study investigates professionals' views and attitudes on facilitating and hindering factors of implementing client-oriented health promotion programs and thus will provide a solid basis for future research activities and evaluation studies in the field of health promotion implementation.

ELIGIBILITY:
Inclusion Criteria:

* Professionals from different levels of the organizational hierarchies
* Professionals from different professional groups
* Professionals with preferably differing views on the usefulness of the health promotion program

Exclusion Criteria:

-

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The aim of this study is to investigate professionals' (teachers', health professionals', care aids') views and attitudes that influence the implementation of client-oriented health promotion programs in organizational settings in Austria. Therefore, 90 professionals will be interviewed: 30 in schools, 30 in hospitals, and 30 in LTC-facilities.
Sampling Method: Non-Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2012-02; Primary Completion 2015-03 (Estimated); Study Completion 2015-03 (Estimated)

PRIMARY OUTCOMES:
Professionals' perspectives towards the implementation process of health promotion programs compositely measured by qualitative semi-structured interviews and non-participant observation | 9 months
  Semi-structured interviews: During different stages of the implementation process, a number of professionals responsible for implementation in each organizational setting are invited for an in-depth interview to gain insight into the implementation of the health promotion program. An interview guide is used to ask participants about the program's content, recruitment, fidelity, and satisfaction with the dissemination strategy, and overall satisfaction with the health promotion program. Facilitators and barriers for implementation, as well as intentions and opportunities for future implementation of health promotion programs are discussed.
  Non-participant observation: In addition, it is observed how professionals across schools, hospitals, and LTC-facilities implement the health promotion program. Non-participant observation is conducted two times in each organizational setting.

SECONDARY OUTCOMES:
Investigation of formal prerequisites of the implementation process measured by extensive document analysis | 9 months
  Documentary data, such as organizational charts or program descriptions of the health promotion programs, are gathered. Therewith, the investigators analyze formal structures and processes within the organizations as well as the formal requirements and goals of the health promotion program.